CLINICAL TRIAL: NCT05120960
Title: A Phase 1a/1b Study to Determine the Recommended Phase 2 Dose, of Tepotinib in Participants With MET Alterations and Brain Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0281; NCI-2021-12845 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — tepotinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): will receive tepotinib alone
  Interventions: Drug: tepotinib
- Group B (Experimental): will receive tepotinib and osimertinib
  Interventions: Drug: tepotinib; Drug: tepotinib plus osimertinib

INTERVENTIONS:
Drug: tepotinib — Given by PO
Drug: tepotinib plus osimertinib — Given by PO
  Arms: Group B

SUMMARY:
This is a single center, multi-arm, biomarker-driven phase 1 study to assess the RP2D, PK/PD, safety, and activity of tepotinib in participants with MET alterations and brain tumors. Eligible patients include those with brain metastases or glioblastoma, including patients who are surgical candidates. In patients with EGFR+ NSCLC with EGFR-TKI resistance and MET amplification, tepotinib will be given in combination with osimertinib. This phase 1 study will be conducted in 2 parts, Phase 1a (dose exploration) and Phase 1b (dose expansion). Phase 1a will include a surgical resection window of opportunity component. Phase 1b (dose expansion) can open once the relevant RP2D has been estimated in Phase 1a (dose exploration). Phase 1a (Dose Exploration): Patients will be assigned to dose levels within a Group as outlined in the Statistical Analysis Plan. Group A will be comprised of patients who are surgical resection candidates with newly-diagnosed or recurrent brain metastases and MET alteration. Group B will be comprised of patients who are surgical resection candidates with recurrent glioblastoma and MET alteration. Group C will be comprised of patients with newly-diagnosed or recurrent brain metastases and epidermal growth factor receptor mutated (EGFR+) non-small cell lung cancer (NSCLC). Phase 1b (Dose Expansion): Upon completion of the Phase 1a (dose exploration) component and estimation of a RP2D, dose expansion may proceed within Group A (consisting of patients with brain metastasis and MET alteration) and Group C (EGFR+ NSCLC brain metastasis, TKI resistance, and MET amplification). Dose expansion in these 2 groups may be done concurrently, but enrollment in each group does not require completion of the entire Phase 1a component of the study. There will not be a Group B (glioblastoma) in Phase 1b. Patients in Phase 1b will not undergo surgical resection.

DETAILED DESCRIPTION:
Phase Ia:

A. To determine the recommended phase II dose (RP2D) of tepotinib for patients with brain metastasis and MET alterations (Group A)

B. To determine RP2D of tepotinib in patients with GLIOBLASTOMA with MET alterations (Group B)

C. To determine RP2D of tepotinib in combination with osimertinib in patients with EGFR+ NSCLC with EGFR TKI resistance and MET amplification (Group C)

Phase 1b:

A. To determine intracranial clinical benefit of tepotinib in brain mets, as measured by RANO-BM, in patients with NSCLC and METex14-skipping mutations (Group A) C. To determine intracranial clinical benefit of tepotinib in combination with osimertinib, in brain metastasis, as measured by RANO-BM, in patients with EGFR+ NSCLC with EGFR TKI resistance and MET amplification (Group C)

2.2 Secondary Objectives:

Phase 1a:

A1. To evaluate the safety and toxicity of tepotinib in treating brain metastasis in patients with MET alterations in Group A, as measured by CTCAE, version 5.0 A2. To evaluate the PK/PD (including phosphomet level) of tepotinib in brain metastasis tissue and CSF in patients with MET alterations in Group A A3. To determine overall survival in Group A A4. To determine progression-free survival for intracranial disease and extracranial disease in Group A A5. To determine intracranial objective response rate according to RANO-BM and the modified Response Evaluation Criteria in Solid Tumors (mRECIST) [Qianet al., 2017] of Group A A6. To determine extracranial objective reponse rate as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 of Group A A7. To identify the site of first progression (intracranial vs extracranial) in Group A A8.To determine the duration of intracranial response by BM-RANO and by mRECIST in Group A A9. To determine the duration of extracranial response by RECIST 1.1 in Group A A10. To determine the time to intracranial progression (defined as progression of existing lesions and development of new lesions) in Group A A11. To explore the patient experience with treatment using patient-reported outcomes (PROs) using the MDASI-BT and EQ-5D-5L questionnaires in Group A A12. To identify the frequency of grade 3+ toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months in Group A A13. To determine changes in dose, duration and frequency of steroid use for symptomatic management in Group A

B1. To evaluate the safety and toxicity of tepotinib in treating glioblastoma in patients with MET alterations (Group B), as measured by CTCAE, version 5.0 B2. To evaluate the PK/PD (including phosphomet level) of tepotinib in glioblastoma tissue and CSF in patients with MET alterations in Group B B3. To determine survival (PFS, OS) of Group B B4. To determine objective response rate according to RANO of Group B B5.To determine the duration of response by RANO in Group B B6. To determine the time to progression (defined as progression of existing lesions and development of new lesions) in Group B B7. To explore the patient experience with treatment using patient-reported outcomes (PROs) using the MDASI-BT and EQ-5D-5L questionnaires in Group B B8. To identify the frequency of grade 3+ toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months in Group B B9. To determine changes in dose, duration and frequency of steroid use for symptomatic management in Group B

C1. To evaluate the safety and toxicity of the combination of osimertinib and tepotinib in treating patients with EGFR+ NSCLC with EGFR TKI resistance and MET amplification, with (Group C), as measured by CTCAE, version 5.0 C2. To evaluate the PK/PD (including phosphomet level) of tepotinib in CSF in patients with EGFR+ NSCLC with EGFR TKI resistance and MET amplification treated with the combination of osimertinib and tepotinib (Group C) C3. To determine overall survival in Group C C4. To determine progression-free survival for intracranial disease and extracranial disease in Group C C5. To determine intracranial objective response rate according to RANO-BM and mRECIST of Group C C6. To determine extracranial objective response rate as assessed by RECIST v1.1 for Group C C7. To identify the site of first progression (intracranial vs extracranial) in Group C C8.To determine the duration of intracranial response by BM-RANO and by mRECIST in Group C C9. To determine the duration of extracranial response by RECIST 1.1 in Group C C10. To determine the time to intracranial progression (defined as progression of existing lesions and development of new lesions) in Group C C11. To explore the patient experience with treatment using patient-reported outcomes (PROs) using the MDASI-BT and EQ-5D-5L questionnaires in Group C C12. To identify the frequency of grade 3+ toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months in Group C C13. To determine changes in dose, duration and frequency of steroid use for symptomatic management in Group C

Phase 1b:

A1. To evaluate the safety and toxicity of tepotinib as measured by CTCAE, version 5.0 in patients with NSCLC and METex14-skipping mutations (Group A) A2. To evaluate the PK/PD (including phosphomet level) of tepotinib in the CSF in patients with NSCLC and METex14-skipping mutations (Group A) A3. To determine overall survival in Group A A4. To determine progression-free survival for intracranial disease and extracranial disease in Group A A5. To determine intracranial objective response rate according to RANO-BM and mRECIST of Group A A6. To determine extracranial objective reponse rate as assessed by RECIST v1.1 of Group A A7. To identify the site of first progression (intracranial vs extracranial) in Group A A8.To determine the duration of intracranial response by BM-RANO and by mRECIST in Group A A9. To determine the duration of extracranial response by RECIST 1.1 in Group A A10. To determine the time to intracranial progression (defined as progression of existing lesions and development of new lesions) in Group A A11. To explore the patient experience with treatment using patient-reported outcomes (PROs) using the MDASI-BT and EQ-5D-5L questionnaires in Group A A12. To identify the frequency of grade 3+ toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months in Group A A13. To determine changes in dose, duration and frequency of steroid use for symptomatic management in Group A

C1. To evaluate the safety andtoxicity as measured by CTCAE, version 5.0, in patients with EGFR+ NSCLC with EGFR TKI resistance and MET amplification (Group C) C2. To evaluate the PK/PD (including phosphomet level) of tepotinib in CSF in patients with EGFR TKI resistance and MET amplification (Group C) C3. To determine overall survival in Group C C4. To determine progression-free survival for intracranial disease and extracranial disease in Group C C5. To determine intracranial objective response rate according to RANO-BM and mRECIST of Group C C6. To determine extracranial objective reponse rate as assessed by RECIST v1.1 for Group C C7. To identify the site of first progression (intracranial vs extracranial) in Group C C8.To determine the duration of intracranial response by BM-RANO and by mRECIST in Group C C9. To determine the duration of extracranial response by RECIST 1.1 in Group C C10. To determine the time to intracranial progression (defined as progression of existing lesions and development of new lesions) in Group C C11. To explore the patient experience with treatment using patient-reported outcomes (PROs) using the MDASI-BT and EQ-5D-5L questionnaires in Group C C12. To identify the frequency of grade 3+ toxicities at 4 weeks, and 3, 6, 9, 12 and 18 months in Group C C13. To determine changes in dose, duration and frequency of steroid use for symptomatic management in Group C

ELIGIBILITY:
Participant Inclusion Criteria:

In order to be eligible for participation in this trial, the participant must:

1. Willing and able to provide written informed consent for the trial.
2. 18 years of age on day of signing informed consent.
3. Performance status of > 60 on the KPS (Karnofsky Performance Status) scale, or ECOG (Eastern Cooperative Oncology Group) performance score of 0 or 1.
4. MRI of the brain consistent with either new or progressive brain metastasis or recurrent glioblastoma.
5. Group A: Histologically-confirmed primary cancer or brain metastasis with MET alteration identified through molecular testing.
6. Group B: Histiologically-confirmed WHO grade IV glioma (glioblastoma or gliosarcoma) with MET alteration identified through molecular testing.

   1. Patients will be eligible if the original histology was low-grade glioma and a subsequent histiological diagnosis of grade IV glioma is made at some point along the disease trajectory.
   2. Note: Patients with IDH wildtype grade III anaplastic astrocytoma (1p19q intact) are also elgibile, as these tumors are expected to behave similarly to grade IV glioma.
   3. At first, second or third recurrence of glioblastoma, and patients must have received prior radiation and/or chemotherapy.
7. Group C: NSCLC with documented activating mutation of the EGFR receptor including T790M status, and with acquired resistance on previous EGFR-TKI therapy, and MET alteration identified through molecular testing.

   a. Patients must have radiological documentation of disease progression on previous EGFR-TKI therapy.

   b. Patients may have received osimertinib. If brain mets progression occurs on osimertinib, patient will be eligible if continues osimertinib.
8. Phase 1b, Group A: Patients must have NSCLC (confirmed by either histology or cytology) with documented METexon14-skipping mutations identified in primary or brain metastasis tissue and/or in circulating tumor DNA in plasma (liquid biopsy).
9. Phase 1a, Groups A and B participants must require surgical resection for clinical care.

   1. Phase 1a, Group A: Patient must be surgical candidate for brain metastasis (solitary met, single met > ~ 2 cm (surgeon's discretion), multiple mets but one large met, symptomatic met controlled on steroid, and/or highly radioresistant met), but not require immediate surgery.
   2. Phase 1a, Group B: Patient must be surgical candidate for glioblastoma, as determined by treating physician, but not require immediate surgery.

2. Phase 1a, Group C and Phase 1b, Groups A and C participants must have small, minimally symptomatic/asymptomatic brain metastasis that do not require surgical resection.

3. Measurable disease

a. Groups A and C: Presence of at least 1 independently verified measurable brain metastasis in accordance with a modified RANO-BM (see Section 6.1.6, Tumor Imaging and Assessment of Disease) that can be accurately assessed at baseline with ≥ 5 mm* in the longest diameter with MRI, which is suitable for accurate repeated measurements and that preferably was not previously irradiated or biopsied *and must be surgical candidate b. Group B: Presence of measurable glioblastoma, per RANO criteria, and that can be accurately assessed at baseline with ≥ 5 mm* in the longest diameter with MRI, which is suitable for accurate repeated measurements *and must be surgical candidate

4. Willing to undergo CSF sampling via lumbar puncture. 5. No medical contraindication to lumbar puncture (to include severe coagulopathy, radiographic concern for impending herniation or obstructive hydrocephalus, or soft tissue infection at puncture site, as outlined in MD Anderson institutional policy).

1. Patient may still enroll but LP may be deferred if at any time the treating physician determines that it would be unsafe to perform this procedure due to the characteristics (size, associated edema, etc) of the brain tumor 6. If taking steroids, stable or decreasing dose of steroids for at least 5 days prior to enrollment; no more than 4 mg dexamethasone (or equivalent) total per day for patients with brain metastasis, and no more than 8 mg per day for patients with glioblastoma.

   7. Demonstrate adequate organ function as defined in Table 1; all screening labs should be performed within 14 days prior to registration (see Table 1).

   Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR
   * 60 mL/min for participant with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

     * 5 X ULN for participants with liver metastases Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   ≤1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ACreatinine clearance should be calculated per institutional standard.

   8. Female patients of childbearing potential should have a negative serum pregnancy test.

   9. Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity, for the course of the study through 28 days after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

   10. Male patients should agree to use an adequate method of contraception starting with the first dose of study therapy through 28 days after the last dose of study therapy.

   11. For patients with brain mets, if patient had prior WBRT or SRS, progression in any measurable brain metastasis must have occurred at least 1 month after the end of radiation therapy.

   12. First day of study drug must be more than 2 weeks from last day of any radiation to the brain or spinal cord/cauda equina.

   13. Patients with minimally symptomatic brain metastases may be enrolled without prior radiation therapy to the brain if they do not require immediate surgical or radiation therapy in the opinion of the treating investigator and in the opinion of a radiation therapy or neurosurgical consultant.

   Participant Exclusion Criteria:

   1. Currently participating in or has participated in a study of an investigational agent (with the exception of participating in which the investigational agent was a 1st, 2nd, or 3rd generation EGFR-TKI) within 4 weeks prior to study enrollment.

   2. Any unresolved toxicity Grade 2 or higher according to NCI-CTCAE version 5, from previous anticancer therapy, with the exception of alopecia. 3. Need for transfusion within 14 days prior to enrollment. 4. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.

   5. Active infection requiring systemic therapy. 6. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

   7. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

   8. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 28 days after the last dose of trial treatment.

   9. History of ILD or interstitial pneumonitis including radiation pneumonitis that required steroid treatment.

   10. Impaired cardiac function:

   - Left ventricular ejection fraction < 45% defined by echocardiography
   * Serious arrhythmia
   * Unstable angina pectoris
   * Congestive Heart Failure New York Heart Association III and IV
   * Myocardial infarction, stroke, or transient ischemic attack within the last 6 months prior to study entry.
   * Corrected QT interval (QTcF) > 470 ms for women and > 450 ms for men at screening.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives, or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.

     11. Hypertension uncontrolled by standard therapies (not stabilized to < 150/90 mmHg).

     12. Group C: Contraindication to the administration of osimertinib. 13. Medical history of liver fibrosis/cirrhosis. 14. Medical history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.

     15. Known human immunodeficiency virus positivity. 16. Group C: Has not received an EGFR-TKI containing treatment prior to enrollment into the study 17. Prior treatment with other agents targeting the HGF/MET pathway such as crizotinib, capmatinib, savolitinib, foretinib, glesatinib, cabozantinib, merestinib, onartuzumab, rilotumumab, emibetuzumab, and ficlatuzumab.

     18. Participants currently receiving (or unable to stop use at least 1 week prior to enrollment) medications or herbal supplements known to be potent inducers of CYP3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
To determine the recommended phase II dose (RP2D) of tepotinib for patients with brain metastasis and MET alterations (Group A) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O'Brien, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org